CLINICAL TRIAL: NCT02338661
Title: Clinical Observation Study With the SBG Stem
Status: Completed | Type: Observational
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: D8319
Record Dates: First submitted 2014-12-12; First posted 2015-01-14 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Arthroplasty, Hip Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: SBG hip stem

SUMMARY:
This study is a prospective, single-center, postmarket clinical observation to observe the clinical and radiographic long-term performance of the SBG hip stem.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring the implantation of the SBG hip stem

Exclusion Criteria:

* general medical contraindications to surgery
* acute or recent infection of joint
* atrophy or deformation of upper femur
* muscular atrophy or neuromuscular disease
* pathologic fractures
* per- and subtrochanteric fractures
* revision of failed hip endoprosthesis
* hypersensitivity to used materials
* any conditions preventing stable anchoring of the hip prosthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2004-01; Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score | Baseline and 10 years post surgery
  Change in Harris Hip Score from Baseline to 10 years post surgery. The Harris Hip Score scales from 0-100 with higher values representing a better score.

SECONDARY OUTCOMES:
Assessment of position of hip stem | Baseline and 10 years post surgery
  Change in hip stem position from Baseline to 10 years post surgery.
Radiographic Analysis: classification of osseointegration of hip stem | 10 years post surgery
Radiographic Analysis: radiolucent lines around hip stem | 10 years post surgery
  Radiographic measurements will be taken of linear radiolucencies. Radiolucent lines will be measured in mm.
Radiographic Analysis: number of participants with femoral osteolysis around hip stem | 10 years post surgery
Radiographic Analysis: bone atrophy around hip stem | 10 years post surgery
  Radiographic measurements will be taken of bone atrophy. Bone atrophy will be measured in mm.
Radiographic Analysis: bone hypertrophy around hip stem | 10 years post surgery
  Radiographic measurements will be taken of bone hypertrophy. Bone hypertrophy will be measured in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Beat Schmid, Dr. med., Principal Investigator — Praxis Klinik Gut Buchs
Locations (1):
- Praxis Klinik Gut Buchs, Buchs, Switzerland